CLINICAL TRIAL: NCT03756220
Title: Combination Therapy of Vitamin C and Thiamine for Septic Shock: Multi-center, Double-blinded, Randomized, Controlled Study
Brief Title: Ascorbic Acid and Thiamine Effect in Septic Shock
Acronym: ATESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tae Gun Shin (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor-Investigator, Tae Gun Shin, Associate professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018R1C1B6006821
Record Dates: First submitted 2018-10-30; First posted 2018-11-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Septic Shock; Sepsis
Keywords: Septic shock; Sepsis; Vitamin C; Thiamine
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Thiamine; Ascorbic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multi-center, Double-blinded, Randomized, Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Combination therapy of vitamin C and thiamine for 2 days.
  Interventions: Drug: Combination therapy of vitamin C and thiamine
- Control (Placebo Comparator): Normal Saline Solution
  Interventions: Drug: Normal saline solution

INTERVENTIONS:
Drug: Combination therapy of vitamin C and thiamine — Vitamin C (50 mg/kg up to 3 g, every 12 hours) and thiamine (200 mg every 12 hours) intravenously administered mixed in 50 mL solution bags of normal saline for 2 days
  Other Names: Ascorbic Acid Injection; Thiamine Injection
  Arms: Treatment
Drug: Normal saline solution — Normal saline solution in a volume to match the treatment components administered mixed in 50 mL solution bags of normal saline for 2 days
  Other Names: 0.9% NaCl
  Arms: Control

SUMMARY:
The aim of this study is to evaluate the efficacy of early metabolic resuscitation with combination therapy using vitamin C and thiamine in improving organ function and survival in patients with septic shock.

DETAILED DESCRIPTION:
Sepsis is a complex disease involving life-threatening organ dysfunction caused by a dysregulated host response to infection and is still associated with unacceptably high mortality. Sepsis management should be undertaken as a medical emergency and focused on timely intervention, including early identification and treatment of infection through appropriate antimicrobial therapy and source control when applicable as well as reversing hemodynamic instability through fluid resuscitation and vasopressor use if necessary. Despite these supportive therapies, morbidity and mortality have remained high, suggesting the need for adjuvant therapies for inflammatory and oxidative stress in patients with sepsis; however, no agents have been proven to definitely improve survival.

Vitamin C plays a role in mediating inflammation through antioxidant activities and is also important as a cofactor/co-substrate for the synthesis of endogenous adrenaline, cortisol, and vasopressin. Recently, several clinical trials have reported the positive effects of vitamin C on outcomes in sepsis or septic shock. During sepsis, vitamin C prevents neutrophil-induced lipid oxidation and protects against the loss of the endothelial barrier. Early intravenous supplementation is therefore needed to limit loss of microcirculation and oxidation of lipids. Thiamine is also a key cofactor for glucose metabolism, the generation of ATP (adenosine triphosphate), and the production of NADPH. Considering acute consumption in the hypermetabolic state, thiamine supplementation might be a reasonable therapeutic adjunct for patients with sepsis and was added to reduce the risk of renal oxalate crystallization. These findings led to a recent before-and-after study showing that treatment of sepsis with a combination of vitamin C, hydrocortisone, and thiamine prevented organ dysfunction and reduced the mortality rate.

The aim of this study is to evaluate the efficacy of early metabolic resuscitation with combination therapy using vitamin C and thiamine in improving organ function and survival in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (> 18 years)
2. Septic shock: sepsis with persisting hypotension requiring vasopressors to maintain a mean arterial pressure ≥65 mm Hg and a serum lactate level >2 mmol/L despite adequate volume resuscitation. Sepsis is defined as clinically suspected or confirmed infection with acute organ failure identified as an acute change in total SOFA score with 2 points or more.

Exclusion Criteria:

1. Transferred patients from other hospitals after application of vasopressors or mechanical ventilation
2. Patients who signed a "Do not attempt resuscitation" order or who had set limitations on invasive care
3. Patients who have a terminal, unresponsive illness and survival discharge is not expected (metastatic terminal cancer, etc.)
4. Patients who experienced cardiac arrest before enrollment or when death is anticipated within 24 hours despite maximal treatment
5. Patients who take more than 1g of Vitamin C per day before enrollment or who take supplemental thiamine
6. Pregnant woman
7. Known Glucose-6-phosphate dehydrogenase deficiency
8. Patients with a history of hypersensitivity to vitamin C or thiamine
9. Known Mediterranean anemia
10. Known hyperoxaluria
11. Known cystinuria
12. Acute gout attack
13. Known oxalate renal stone
14. Patients who meet the inclusion criteria 24 hours after emergency department arrival or when enrollment is delayed more than 24 hours after diagnosis of septic shock
15. Inability or refusal of a subject or legal surrogate to give informed consent

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Delta Sequential Organ Failure Assessment (SOFA) score | Enrollment to 72 hours
  72-hour change in SOFA score, which reflected recovery from organ failure (delta SOFA = SOFA at enrollment - SOFA after 72 hours)

SECONDARY OUTCOMES:
28-day mortality | Day 28
  The number of participants who did not survive until Day 28 will be compared between the treatment and the control group
7-day mortality (early death) | Day 7
  The number of participants who did not survive until Day 7 will be compared between the treatment and the control group
90-day mortality | Day 90
  The number of participants who did not survive until Day 90 will be compared between the treatment and the control group
Time to death | Enrollment to Day 28
  Days until death
In-hospital death | Up to 12 weeks
  The number of participants who did not survive at hospital discharge will be compared between the treatment and the control group
Intensive care unit death (ICU) death | Up to 12 weeks
  The number of participants who did not survive at ICU discharge from the first index ICU admission will be compared between the treatment and the control group
Time to Shock reversal | Enrollment to Day 14
  Days from enrollment to shock reversal until Day 14. Shock reversal is defined as discontinuation of all vasopressors and mean arterial pressure is maintained at 60 mmHg or more for more than 24 hours.
Vasopressor free days | Enrollment to Day 14
  Days not receiving any vasopressor
Ventilator free days | Enrollment to Day 14
  Days not receiving mechanical ventilation
Ventilator duration | Up to 12 weeks
  Days receiving mechanical ventilation during hospital stay
Renal replacement therapy (RRT) free days | Enrollment to Day 14
  Days not receiving Renal replacement therapy
New use of renal replacement therapy (RRT) | Up to 12 weeks
  The number of participants who receive RRT during hospital stay will be compared between the treatment and the control group
New onset or aggravation of acute kidney injury (AKI) | Enrollment to Day 14
  The number of participants who suffer from new onset or aggravation of AKI will be compared between the treatment and the control group
Length of ICU stay | Up to 12 weeks
  Number of days in the ICU during hospital admission
ICU free day | Enrollment to Day 14
  Days not being in the ICU
Length of hospital stay | Up to 12 weeks
  Number of days in the hospital during hospital admission

OTHER OUTCOMES:
CRP (C-reactive protein) change during initial 72 hours | Enrollment to 72 hours
  72-hour change in CRP (%)
Procalcitonin change during initial 72 hours | Enrollment to 72 hours
  72-hour change in procalcitonin (%)
Dose of vasopressor at 24-hour | Enrollment to 24 hours
  Norepinephrine equivalent dose at 24 hours from enrollment
Dose of vasopressor at 48-hour | Enrollment to 48 hours
  Norepinephrine equivalent dose at 48 hours from enrollment
Dose of vasopressor at 72-hour | Enrollment to 72 hours
  Norepinephrine equivalent dose at 72 hours from enrollment
Maximum dose of vasopressor during initial 72 hours | Enrollment to 72 hours
  Maximum norepinephrine equivalent dose during initial 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tae Gun Shin, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (6):
- South Korea (6):
  - Department of Emergency Medicine, Seoul National University Bundang Hospital,, Seongnam-si, Gyeonggi-do
  - Department of Emergency Medicine, Borame Medical Center, Seoul National University, College of Medicine, Seoul
  - Department of Emergency Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine,, Seoul
  - Department of Emergency Medicine, Seoul National University College of Medicine,, Seoul
  - Department of Emergency Medicine, University of Ulsan College of Medicine, Asan Medical Center,, Seoul
  - Department of Emergency Medicine, Yonsei University College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Background] Teng J, Pourmand A, Mazer-Amirshahi M. Vitamin C: The next step in sepsis management? J Crit Care. 2018 Feb;43:230-234. doi: 10.1016/j.jcrc.2017.09.031. Epub 2017 Sep 18. PMID 28934705
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Background] Oudemans-van Straaten HM, Spoelstra-de Man AM, de Waard MC. Vitamin C revisited. Crit Care. 2014 Aug 6;18(4):460. doi: 10.1186/s13054-014-0460-x. PMID 25185110
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Background] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] May JM, Harrison FE. Role of vitamin C in the function of the vascular endothelium. Antioxid Redox Signal. 2013 Dec 10;19(17):2068-83. doi: 10.1089/ars.2013.5205. Epub 2013 May 29. PMID 23581713
- [Background] Leite HP, de Lima LF. Metabolic resuscitation in sepsis: a necessary step beyond the hemodynamic? J Thorac Dis. 2016 Jul;8(7):E552-7. doi: 10.21037/jtd.2016.05.37. PMID 27501325
- [Background] de Grooth HJ, Geenen IL, Girbes AR, Vincent JL, Parienti JJ, Oudemans-van Straaten HM. SOFA and mortality endpoints in randomized controlled trials: a systematic review and meta-regression analysis. Crit Care. 2017 Feb 24;21(1):38. doi: 10.1186/s13054-017-1609-1. PMID 28231816
- [Derived] Park JE, Jo YH, Hwang SY, Kim WY, Ryoo SM, Jang DH, Kim T, Kim YJ, Kim S, Cho H, Lee GT, Chung SP, Choi SH, Shin TG, Suh GJ; Korean Shock Society (KoSS) Investigators. Biomarker Analysis for Combination Therapy of Vitamin C and Thiamine in Septic Shock: A Post-Hoc Study of the ATESS Trial. Shock. 2022 Jan 1;57(1):81-87. doi: 10.1097/SHK.0000000000001850. PMID 34482319
- [Derived] Hwang SY, Park JE, Jo IJ, Kim S, Chung SP, Kong T, Shin J, Lee HJ, You KM, Jo YH, Kim D, Suh GJ, Kim T, Kim WY, Kim YJ, Ryoo SM, Choi SH, Shin TG; Korean Shock Society (KoSS) Investigators. Combination therapy of vitamin C and thiamine for septic shock in a multicentre, double-blind, randomized, controlled study (ATESS): study protocol for a randomized controlled trial. Trials. 2019 Jul 11;20(1):420. doi: 10.1186/s13063-019-3542-x. PMID 31296251